CLINICAL TRIAL: NCT04934410
Title: Induction Agent and Incidence of Hypotension in Heart Failure Patients Undergoing LVAD-Implantation
Acronym: INTENS
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Heidelberg University (Other)
Responsible Party: Principal Investigator, Dr. Adrian Stephan, Principal Investigator, Heidelberg University
Other Study IDs: S-602/2020
Record Dates: First submitted 2021-01-29; First posted 2021-06-22 (Actual); Last update posted 2021-10-19 (Actual); Status verified 2021-10

CONDITIONS: Blood Pressure, Low
Keywords: Blood Pressure; Catecholamines; Heart failure; High risk patients; Left ventricular assist device
MeSH Terms: conditions — Hypotension; Heart Failure | interventions — Etomidate; Midazolam; Sevoflurane

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes

GROUPS / COHORTS (3):
- Patients undergoing Implantation of left ventricular assist device (Etomidate): High-risk heart-failure patients undergoing the implantation of a left ventricular assist device (LVAD). The induction agent is etomidate.
  Interventions: Drug: Etomidate
- Patients undergoing Implantation of left ventricular assist device (Midazolam): High-risk heart-failure patients undergoing the implantation of a left ventricular assist device (LVAD). The induction agent is midazolam.
  Interventions: Drug: Midazolam
- Patients undergoing Implantation of left ventricular assist device (Sevoflurane): High-risk heart-failure patients undergoing the implantation of a left ventricular assist device (LVAD). The induction agent is sevoflurane.
  Interventions: Drug: Sevoflurane

INTERVENTIONS:
Drug: Etomidate — Use of etomidate during induction as decided by attending anesthesiologist
  Groups: Patients undergoing Implantation of left ventricular assist device (Etomidate)
Drug: Midazolam — Use of midazolam during induction as decided by attending anesthesiologist
  Groups: Patients undergoing Implantation of left ventricular assist device (Midazolam)
Drug: Sevoflurane — Use of sevoflurane during induction as decided by attending anesthesiologist
  Groups: Patients undergoing Implantation of left ventricular assist device (Sevoflurane)

SUMMARY:
The induction of anesthesia is one of the most critical situations for high-risk-patients undergoing major surgery. For several reasons, it is crucial to maintain adequate blood pressure and cardiac output during this phase.

This observational study aims to find out if the choice of the induction agent has a major impact on blood pressure and the use of antihypotensive drugs during the induction and the surgical procedure in heart-failure patients undergoing the implantation of a left ventricular assist device (LVAD).

ELIGIBILITY:
Inclusion Criteria:

- Heart failure patients scheduled for implantation of left ventricular assist device (LVAD)

Exclusion Criteria:

* Pregnancy
* Presence of another cardiac assist device in the patient (for example ECLS)
* No consent of the patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with terminal heart failure which are scheduled for implantation of a left ventricular assist device (LVAD)
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2021-11-01 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Post-Induction hypotension | First 30 minutes after induction of anesthesia
  The incidence of hypotension in the first 30 minutes after the induction of anesthesia

SECONDARY OUTCOMES:
Antihypotensive drugs after induction | First 30 minutes after induction of anesthesia
  Use of antihypotensive drugs during the first 30 minutes after induction of anesthesia
Antihypotensive drugs during the procedure | Begin of the procedure until end of the procedure
  Use of antihypotensive drugs during the procedure
Length of stay on the intensive care unit (ICU) | After the procedure and transport to intensive care unit, total time in hours until submission from I. Expected time frame is 48 to 96 hours.CU
  The time the patient has to be treated on intensive care unit after the procedure (in hours) before submission.
Delirium | First 24 hours after the end of the procedure
  Diagnosis of postoperative delirium
Kidney | First 28 days after procedure
  Occurrence of acute kidney failure as defined by Kidney Disease: Improving Global Outcomes (KDIGO)
Mortality | First 28 days after procedure
  Mortalitiy in the first 28 days after the procedure

CONTACTS AND LOCATIONS:
Overall Officials: Adrian E Stephan, MD, Study Director — Department of Anesthesiology, Heidelberg University Hospital, Heidelberg, Germany